CLINICAL TRIAL: NCT01413750
Title: Phase II Randomized Study of Vorinostat or Placebo in Combination With Carboplatin and Paclitaxel for Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Carboplatin and Paclitaxel With or Without Vorinostat in Treating Patients With Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: CTEP Initiated Action
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NCI-2010-02203; NCI-2010-02203 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-102 (Other: City of Hope Comprehensive Cancer Center); 8703 (Other: CTEP); N01CM00038 (NIH); N01CM00071 (NIH); N01CM00100 (NIH); N01CM62209 (NIH); P30CA033572 (NIH); U01CA099168 (NIH)
Record Dates: First submitted 2011-08-05; First posted 2011-08-10 (Estimated); Results first posted 2015-08-18 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-10

CONDITIONS: Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: interventions — Carboplatin; Paclitaxel; Taxes; Vorinostat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Arm I (paclitaxel, carboplatin, vorinostat) (Experimental): Patients receive paclitaxel IV over 3 hours, and carboplatin IV over 30 minutes on day 0. Patients also receive vorinostat PO once daily on days -2 to 2.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Drug: Vorinostat
- Arm II (paclitaxel, carboplatin, placebo) (Active Comparator): Patients receive paclitaxel and carboplatin as in arm I. Patients also receive placebo PO once daily on days -2 to 2.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Other: Placebo Administration

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Placebo Administration — Given PO
  Arms: Arm II (paclitaxel, carboplatin, placebo)
Drug: Vorinostat — Given PO
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza
  Arms: Arm I (paclitaxel, carboplatin, vorinostat)

SUMMARY:
Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Vorinostat may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether giving carboplatin and paclitaxel together is more effective with or without vorinostat in treating non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare progression-free survival associated with the combination of carboplatin, paclitaxel and vorinostat versus carboplatin, paclitaxel and placebo for patients with previously untreated, advanced NSCLC.

SECONDARY OBJECTIVES:

I. To determine the response rate, time to treatment failure, and overall survival for the two regimens.

II. To assess the safety profile of the regimen of vorinostat, carboplatin and paclitaxel for patients with advanced NSCLC.

III. To understand the mechanistic aspects of drug effect by conducting correlative science studies on peripheral blood and archived tumor tissue.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive paclitaxel IV over 3 hours, and carboplatin IV over 30 minutes on day 0. Patients also receive vorinostat orally (PO) once daily on days -2 to 2.

ARM II: Patients receive paclitaxel and carboplatin as in arm I. Patients also receive placebo PO once daily on days -2 to 2.

In both arms, treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, quarterly for 1 year, and then twice a year thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed non-small cell lung cancer
* No prior chemotherapy for advanced or metastatic disease
* ECOG performance status 0 or 1
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral CT scan
* Life expectancy of greater than 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy in a metastatic setting
* Patients may not be receiving any other investigational agents
* Patients with untreated brain metastases should be excluded from this clinical trial; however, patients who have stable brain disease (should be off corticosteroids) at least 3 weeks after completion of appropriate therapy are eligible
* Patients who have received any prior HDAC inhibitor (except valproic acid for seizure control provided that the valproic acid has been stopped at least 30 days before beginning therapy on this protocol) are excluded from this study
* Peripheral neuropathy of severity greater than grade 1
* Known history of allergic reactions to paclitaxel
* Prior therapy with paclitaxel
* Inability to take oral medications on a continuous basis; patients unable to swallow the vorinostat capsules whole are ineligible (the capsules cannot be crushed or broken)
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with vorinostat; women of childbearing potential must use an appropriate double barrier method of birth control (such as female use of a diaphragm, intrauterine device [IUD], sponge and spermicide, in addition to the male use of a condom) or a prescribed birth control implant or practice abstinence; both double barrier contraception and implants must be used for at least one week prior to the start of the research study and continue for at least two weeks following the last study visit; please note that birth control pills should not be used while on this study as they may have a negative interaction with the experimental drug in this study
* HIV-positive patients receiving combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2010-11-08 (Actual); Primary Completion 2013-04-14 (Actual); Study Completion 2013-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chandra P Belani, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (13):
- United States (13):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Dose Level 1: Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients also receive 600 mg QD of Vorinostat on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Vorinostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Phase I: Dose Level 2: Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients also receive 800 mg QD of Vorinostat on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Vorinostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Phase II: Vorinostat: Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients randomized to 800 mg QD of Vorinostat on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Vorinostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Phase II: Placebo: Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients randomized to placebo on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Placebo: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II: Vorinostat | Phase II: Placebo
Started | 6 | 6 | 4 | 7
Completed | 6 | 6 | 4 | 7
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase II (Vorinostat): Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients randomized to 800 mg QD of Vorinostat on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Vorinostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Phase II (Placebo): Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients randomized to 800 mg QD of Vorinostat on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Placebo: Given PO
  Laboratory Biomarker Analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II (Vorinostat) | Phase II (Placebo) | Total
Number analyzed (Participants) | 6 | 6 | 4 | 7 | 23
Age, Continuous [Median (Full Range); unit: years] | 61 [53 to 64] | 59 [24 to 79] | 72 [62 to 77] | 65 [52 to 72] | 63 [24 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 7
  Male | 4 | 4 | 3 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 4 | 7 | 23

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Estimated using the product-limit method of Kaplan and Meier.
  PFS defined as time from randomization to progression or death due to any cause.
  Progression defined as Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first day of treatment to the first observation of disease progression or death due to any cause, assessed up to 1 year
Population: Due to early termination phase II portion of the study did not reach planned accrual.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II: Vorinostat | Phase II: Placebo
Number analyzed (Participants) | 4 | 7
months | 4.1 [0.5 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 7.3 [0.4 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

2. Secondary Outcome: Dose Limiting Toxicity (DLT) (Phase I)
Description: DLT is defined as any grade III or higher non-hematological toxicity except nausea, vomiting or alopecia. Nausea or vomiting (> grade 2) that last longer than 48 hours despite maximal medical therapy. Absolute neutrophil count < 1000/uL lasting longer than 7 days. Grade 4 thrombocytopenia (platelet < 25,000/uL). Grade 3 or 4 neutropenia associated with sepsis or fever > 38 C. Delay in starting cycle 2 by more than 2 weeks due to toxicity.Abnormal non-hematological laboratory criteria (Grade 3 or higher) will be considered a DLT, if clinically significant and drug-related. If baseline value is elevated prior to drug therapy, an increase will not be considered a DLT unless there is an elevation by more than 2 grades, and it is of clinical significance. Dose escalation schedule for vorinostat: 600 mg QD; 800 mg QD.
Time Frame: 4 weeks from start of treatment, up to 1 year
Measure: Number; unit: participants with DLTs
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2
Number analyzed (Participants) | 6 | 6
participants with DLTs | 1 | 0

3. Secondary Outcome: Maximum Tolerated Dose (MTD) (Phase I)
Description: The highest dose tested in which fewer than 33% of patients experience an attributable DLT to the study drug, when at least 6 patients are treated at that dose and are evaluable for toxicity. The MTD is one dose level below the lowest dose in which 33% or more of the patients experience a DLT. The MTD is based on the first cycle of therapy. The recommended Phase II dose is generally the MTD, although secondary considerations of toxicity and dose reductions on subsequent cycles and other secondary considerations may result in the recommended Phase II dose being below the MTD.
Time Frame: 4 weeks from start of treatment, up to 1 year
Measure: Number; unit: mg
Groups:
- Phase I: All patients enrolled on the Phase I (safety lead-in) portion of the study.
Arm/Group | Phase I
Number analyzed (Participants) | 12
mg | 800

ADVERSE EVENTS:
Time Frame: Adverse events collected over a period of 2 years and 4 months
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Groups:
- Phase II: Vorinostat: Patients receive A fixed dose of Carboplatin at AUC 6 mg/ml.min iv on day 0 of each cycle and Paclitaxel 200 mg/m2, iv on day 0 of each cycle. Patients randomized to 800 mg QD of Vorinostat on days -2 to 2. Each cycle is 21 days.
  Paclitaxel: Given IV
  Carboplatin: Given IV
  Voninostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Arm/Group | Phase I: Dose Level 1 | Phase I: Dose Level 2 | Phase II: Vorinostat | Phase II: Placebo
Serious Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 3/4 | 5/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 1 (N=6) | Phase I: Dose Level 2 (N=6) | Phase II: Vorinostat (N=4) | Phase II: Placebo (N=7)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Esophageal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sudden death NOS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 3 (3) | 2 (2) | 2 (3) | 4 (7)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Dose Level 1 (N=6) | Phase I: Dose Level 2 (N=6) | Phase II: Vorinostat (N=4) | Phase II: Placebo (N=7)
Anemia (Blood and lymphatic system disorders) | 5 (20) | 5 (11) | 2 (14) | 6 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (8) | 0 (0) | 0 (0) | 2 (4)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 2 (4) | 2 (4) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 4 (12) | 5 (8) | 2 (7) | 6 (22)
Fever (General disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (4) | 3 (3) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 3 (5) | 1 (2) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 1 (2) | 1 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 2 (4) | 1 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 1 (1) | 1 (2) | 1 (1)
Cardiac troponin I increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Creatinine increased (Investigations) | 1 (1) | 2 (2) | 2 (5) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (12) | 1 (2) | 1 (5) | 3 (8)
Lymphocyte count increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 6 (13) | 2 (3) | 2 (6) | 4 (10)
Platelet count decreased (Investigations) | 3 (5) | 3 (3) | 2 (10) | 4 (11)
Weight gain (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (3) | 1 (1) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 6 (17) | 3 (3) | 2 (12) | 4 (15)
Anorexia (Metabolism and nutrition disorders) | 4 (6) | 2 (2) | 1 (2) | 3 (8)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (5) | 2 (5) | 0 (0) | 3 (6)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (11) | 1 (1) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 1 (2) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (6) | 2 (2) | 0 (0) | 1 (2)
Hyponatremia (Metabolism and nutrition disorders) | 5 (8) | 3 (4) | 2 (3) | 3 (7)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 2 (4) | 2 (7)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (7)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (3) | 1 (2) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (4) | 2 (3)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2) | 1 (2) | 2 (5) | 3 (15)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (6)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (16)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (4) | 4 (5) | 3 (5) | 3 (6)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 3 (3) | 3 (7) | 3 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (9) | 1 (1) | 0 (0) | 2 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (9)
Phlebitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated early by NCI due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less